CLINICAL TRIAL: NCT03034265
Title: Identification of New Biomarkers for the Classification and Monitoring of Difficult-to-treat Arterial Hypertension: Prospective Observational Study
Brief Title: New Biomarkers and Difficult-to-treat Hypertension
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Study 3003
Record Dates: First submitted 2017-01-19; First posted 2017-01-27 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
Keywords: hypertension; exosome; angiotensin; sodium channel; kidney; aldosterone; renin; urine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the concentrations and variabilities of urinary exosomal sodium channels and plasma angiotensins in patients with difficult-to-treat arterial hypertension and to investigate their dependency on clinical parameters and sampling conditions.

DETAILED DESCRIPTION:
Background:

Difficult-to-treat hypertension is characterized by uncontrolled blood pressure despite 2 or more antihypertensive drugs. In many cases, abnormal renal Na and volume handling plays a central role. Arterial vasoconstriction and renal function are regulated by the renin-angiotensin-aldosterone system (RAAS) and its effector hormones angiotensin II and aldosterone. Both control renal tubular function and Na excretion. Blocking the renin-angiotensin-system pharmacologically is therefore a current standard approach to treat hypertension. However, there is great clinical need to improve the classification of hypertensive patients and to predict patient sensitivity to different therapeutic strategies more precisely by new biomarkers that take into account tubular function and the various bioactive angiotensin fragments.

Ang fragments generated by non-canonical enzymatic pathways such as Ang III co-exist with Ang I and Ang II in plasma. Their profile could help classify hypertensive patients with greater precision than plasma renin and aldosterone alone. Furthermore, urinary exosomes are small membrane vesicles (<0.1 μm) shed into the urine by tubular epithelial cells. They contain tubular Na channels known as targets of furosemide and thiazide drugs used to treat volume overload and arterial hypertension. Na channel concentrations in the tubules are regulated by Ang II and aldosterone. Exosomal Na channel abundance could thus give valuable extra information on the actual tubular functional status not provided by standard laboratory tests of plasma renin and aldosterone or urinary electrolytes alone. Plasma Ang peptide profiles and urinary exosomal Na channels could improve the classification of patients with difficult-to-control hypertension and inform antihypertensive treatment decisions. The usual concentrations and variabilities of these biomarkers are a prerequisite for the planning of future validation studies. However, data are still lacking in this population.

Study aim:

This study aims to determine the concentration and interindividual variability of urinary exosomal sodium channels and of plasma angiotensins (candidate biomarkers) in patients with difficult-to-treat arterial hypertension and to determine their dependency on sampling conditions, dietary salt intake, and plasma renin and aldosterone concentrations.

Candidate biomarker definition:

* Plasma Ang peptides planned for determination in the study are Ang I and II and its metabolites Ang 2-10, 2-8, 3-8, 1-7, 2-7, 3-7, 1-5 (Ang peptide profile).
* Urinary exosomal Na channel proteins planned for determination are Na+-Cl- cotransporter (NCC), epithelial sodium channel (ENaC) subunits and Na-K-Cl cotransporter type 2 (NKCC 2).

Study type:

This is an investigator initiated, monocentric observational pilot study in 24 ambulatory patients with difficult-to-treat hypertension who meet the inclusion criteria and none of the exclusion criteria.

Setting:

The study is performed at the outpatient hypertension clinic of the University clinic for nephrology, hypertension and clinical pharmacology, Inselspital, Bern University Hospital, Bern, Switzerland.

Objectives:

* The primary objective of the study is to determine the concentration and interindividual variability of urinary exosomal Na channels and of plasma angiotensin peptides under standardized clinical sampling conditions in patients with difficult-to-treat hypertension.
* The secondary objectives of the study are

  1. to determine the association of these candidate biomarkers with urinary Na excretion, plasma renin and aldosterone concentrations, and aldosterone-to-renin ratios on clinical visit 2,
  2. to assess the repeatability of biomarker determinations under spontaneous (visit 1) compared to standardized sampling conditions (visit 2).

Study plan and procedures:

The concentrations of the candidate biomarkers are determined in blood and spot urinary samples obtained on the first clinical visit (visit 1) and again under standardized laboratory conditions on the second clinical visit (visit 2) scheduled 5-31 days later and after stopping RAAS inhibitory drugs, beta-adrenoceptor blockers, centrally acting antihypertensives and diuretics for an appropriate period, as necessary. Ca-antagonists and alpha-adrenoceptor blockers are allowed to treat hypertension.

Determinations of candidate biomarkers are made in parallel with clinical blood and urine tests performed routinely. On visit 2, these tests include supine and standing plasma renin and aldosterone measurements under standardized conditions in the morning after 1 h rest and again after 1 hour walking .

Biological samples are processed according to standardized laboratory protocols. Plasma Ang peptides are determined by gas chromatography-mass spectrometry. Urinary exosomal proteins are determined by Western-Blot using specific antibodies. Blood concentrations of antihypertensive drugs are determined by liquid chromatography mass spectrometry to analyze medication use and adherence on visits 1 and 2. Clinical data and routine laboratory results for visits 1 and 2 are obtained from patient files.

Recruitment of participants: consecutive ongoing participant recruitment is performed in daily clinic practice by the investigators who check referrals for potential eligibility.

Participation: study participation begins with study inclusion on visit 1 and ends with completion of visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥2 antihypertensive drugs for ≥3 months
* Reported blood pressure ≥140/90 mmHg and/or patient reported as having medically uncontrolled hypertension by the referring physician
* Age ≥18 years, capacity to provide and granted written informed consent

Exclusion Criteria:

* Chronic stage 4-5 renal insufficiency; glomerulonephritis, liver insufficiency (Child-Pugh B or C), chronic obstructive pulmonary disease Global Initiative for Obstructive Lung Disease grade 4; chronic heart failure New York Heart Association class IV
* Known secondary hypertension
* Mandatory RAAS-blockers (e.g. converting enzyme inhibitors, angiotensin type 1 receptor blockers), beta-adrenoceptor blockers, centrally acting sympatholytics and diuretics that cannot be paused adequately before visit 2
* Mean sitting office blood pressure >190/110 mmHg measured 3x on visit 1
* Normotension on visit 1 (mean seated office blood pressure measured 3x <140/90 mmHg)
* Insufficient knowledge of project language and absence of an interpreter for study communications
* Pregnancy or lactation
* Scheduled clinical visit 2 outside routine workflow time-line (<5 or >31 days after visit 1)
* Inability to follow procedures (e.g. relevant psychiatric disorder or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Amblatory patients with difficult-to-treat hypertension referred to the hypertension clinic for evaluation
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Ang peptides | 2nd scheduled visit (5 days to 4 weeks after 1st visit)
Urinary concentration of exosomal Na channel proteins | 2nd scheduled visit (5 days to 4 weeks after 1st visit)

SECONDARY OUTCOMES:
24h urinary Na excretion | 2nd scheduled visit (5 days to 4 weeks after 1st visit)
Plasma renin concentration | 2nd scheduled visit (5 days to 4 weeks after 1st visit)
Plasma aldosterone concentration | 2nd scheduled visit (5 days to 4 weeks after 1st visit)
Repeatability of Ang peptide and urinary exosomal Na channel concentrations under spontaneous vs. standardized laboratory conditions. | 1st visit vs. 2nd scheduled visit (5 days to 4 weeks after 1st visit)
  Statistical agreement is tested.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Bohlender, M.D., Principal Investigator — Inselspital, Bern University Hospital, Freiburgstr. 4, 3010 Bern, Switzerland
Locations (1):
- Department of Nephrology and Hypertension, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Interested third parties may have access to project data by contacting the leading investigator. Only anonymous data are shared, also in case with third parties with lower data protection standards than Swiss or European Union, to safeguard confidentiality.

REFERENCES:
- [Background] Campbell DJ, Nussberger J, Stowasser M, Danser AH, Morganti A, Frandsen E, Menard J. Activity assays and immunoassays for plasma Renin and prorenin: information provided and precautions necessary for accurate measurement. Clin Chem. 2009 May;55(5):867-77. doi: 10.1373/clinchem.2008.118000. Epub 2009 Mar 5. PMID 19264850
- [Background] Egan BM, Zhao Y, Axon RN, Brzezinski WA, Ferdinand KC. Uncontrolled and apparent treatment resistant hypertension in the United States, 1988 to 2008. Circulation. 2011 Aug 30;124(9):1046-58. doi: 10.1161/CIRCULATIONAHA.111.030189. Epub 2011 Aug 8. PMID 21824920
- [Background] Glicklich D, Frishman WH. Drug therapy of apparent treatment-resistant hypertension: focus on mineralocorticoid receptor antagonists. Drugs. 2015 Apr;75(5):473-85. doi: 10.1007/s40265-015-0372-3. PMID 25787734
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] Pisitkun T, Shen RF, Knepper MA. Identification and proteomic profiling of exosomes in human urine. Proc Natl Acad Sci U S A. 2004 Sep 7;101(36):13368-73. doi: 10.1073/pnas.0403453101. Epub 2004 Aug 23. PMID 15326289
- [Background] Te Riet L, van Esch JH, Roks AJ, van den Meiracker AH, Danser AH. Hypertension: renin-angiotensin-aldosterone system alterations. Circ Res. 2015 Mar 13;116(6):960-75. doi: 10.1161/CIRCRESAHA.116.303587. PMID 25767283
- [Background] van der Lubbe N, Jansen PM, Salih M, Fenton RA, van den Meiracker AH, Danser AH, Zietse R, Hoorn EJ. The phosphorylated sodium chloride cotransporter in urinary exosomes is superior to prostasin as a marker for aldosteronism. Hypertension. 2012 Sep;60(3):741-8. doi: 10.1161/HYPERTENSIONAHA.112.198135. Epub 2012 Jul 30. PMID 22851731
- [Background] Wolley MJ, Stowasser M. Resistant Hypertension and Chronic Kidney Disease: a Dangerous Liaison. Curr Hypertens Rep. 2016 Apr;18(5):36. doi: 10.1007/s11906-016-0641-x. PMID 27072829